CLINICAL TRIAL: NCT03978793
Title: MyTPill: A Novel Strategy to Monitor Antiretroviral Adherence Among HIV+ Prescription Opioid Users
Acronym: MyTPill
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: University of Miami (Other); The Miriam Hospital (Other); Massachusetts General Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH); Florida International University (Other)
Responsible Party: Principal Investigator, Edward Boyer, Professor, Ohio State University
Other Study IDs: 2021X0070; R01DA047236 (NIH); K24DA037109 (NIH)
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-05

CONDITIONS: HIV-positive Individuals

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MyTPill: Participants receive digital pills for three months, have a 2-week washout, then switch to Wisepill.
  Interventions: Device: MyTPill, a digital pill

INTERVENTIONS:
Device: MyTPill, a digital pill — MyTPill is a digital pill containing an approved medication
  Other Names: Wisepill, a digital pillbox

SUMMARY:
This study compares several different antiretroviral adherence measures, including digital pills, in HIV+ individuals who are maintained on opioid analgesics.

DETAILED DESCRIPTION:
This study compares digital pills, electronic pill bottles, self-report, and dried blood spots, in measuring adherence to antiretroviral medications containing emtricitabine and tenofovir.

ELIGIBILITY:
Inclusion Criteria:

* HIV+, Viral load >200copies/mL, on single pill containing TDF/FTC, receiving prescription for opioid analgesics

Exclusion Criteria:

* Severe renal or hepatic disease
* Hypersensitivity to silver, magnesium, or zinc following oral use
* Pregnancy
* non-English speaking
* History of Crohn's disease or Ulcerative Colitis
* History of bowel surgery, gastric bypass, or bowel stricture
* History of gastrointestinal malignancy or radiation to the abdomen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV+
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Dried blood spots | six months
  Measurement of dried blood spots for TDF/FTC concentrations
Adherence per two different electronic adherence measures | Six months
  Secondary outcomes are the identification of multi-level factors that are prevalent in the target population most closely linked to ART non-adherence and EAM non-adherence.

SECONDARY OUTCOMES:
Pill counts | Six months
  Count numbers of antiretroviral pills at followup sessions

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Boyer, MD PhD, Principal Investigator — Ohio State University
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bischof JJ, Chai P, Mohamed Y, Padappayil R, Merchant RC, Boyer EW, Rosen R, Reyes-Gibby CC, Viamonte M, W Carrico A. MyTPill: study protocol for a cross-over randomised controlled trial comparing novel strategies to monitor antiretroviral adherence among HIV+ prescription opioid users. BMJ Open. 2023 Jan 10;13(1):e062805. doi: 10.1136/bmjopen-2022-062805. PMID 36627157